CLINICAL TRIAL: NCT02952482
Title: Newborn Screening for Adrenoleukodystrophy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201603025RIND
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2017-07

CONDITIONS: Adrenoleukodystrophy
Keywords: adrenoleukodystrophy; C26:0-lyso-PC
MeSH Terms: conditions — Adrenoleukodystrophy | interventions — ATP Binding Cassette Transporter, Subfamily D, Member 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- newborns testing for ALD: newborns testing for ALD
  Interventions: Procedure: newborns testing for ALD

INTERVENTIONS:
Procedure: newborns testing for ALD — Routine newborn screening dried blood spots sample is used to test if elevation of C26:0-lyso-PC

SUMMARY:
To test if the routine newborn screening dried blood spots can be used to test if elevation of C26:0 lysophosphatidylcholine (C26:0-lyso-PC), a status indicating adrenoleukodystrophy (ALD)

DETAILED DESCRIPTION:
Parents of newborns will be invited to test if their newborns are affected with ALD. The routine newborn screening dried blood spots sample will be used to test the concentration of C26:0-lyso-PC . If positive of a screening test, further confirmation tests including physical examination and other methodology for ALD confirmation will be provided. Genetic counseling and treatment option will be provided, too.

ELIGIBILITY:
Inclusion Criteria:

* Babies born in Taiwan receive regular newborn screening suggested by Ministry of Heath and Welfare.
* Parents or Legal Guardian sign in the informed consent form.

Exclusion Criteria:

* Parents or Legal Guardian do not agree to sign in the informed consent form.

Ages: 2 Days to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: newborns whose parents agree to be tested
Sampling Method: Non-Probability Sample
Enrollment: 45796 (Actual)
Dates: Start 2016-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
numbers of newborn with ALD | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No